CLINICAL TRIAL: NCT06588283
Title: Efficacy and Safety of Ixekizumab or Ixekizumab Concomitantly Administered With Tirzepatide in Adult Participants With Moderate-to-Severe Plaque Psoriasis and Obesity or Overweight: A Phase 3b, Randomized, Multicenter, Open-Label Study (TOGETHER-PsO)
Brief Title: Ixekizumab Concomitantly Administered With Tirzepatide in Adults With Moderate-to-Severe Plaque Psoriasis and Obesity or Overweight
Acronym: TOGETHER-PsO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27243; I1F-MC-RHDC (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis; Obesity
MeSH Terms: conditions — Psoriasis; Obesity | interventions — ixekizumab; Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixekizumab (Experimental): Ixekizumab administered subcutaneous (SC).
  Interventions: Drug: Ixekizumab
- Ixekizumab and Tirzepatide (Experimental): Ixekizumab concomitantly administered with tirzepatide SC.
  Interventions: Drug: Ixekizumab; Drug: Tirzepatide

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
Drug: Tirzepatide — Administered SC.
  Other Names: LY3298176
  Arms: Ixekizumab and Tirzepatide

SUMMARY:
The main purpose of this study is to demonstrate that when participants with moderate to severe plaque psoriasis and obesity or overweight in the presence of at least 1 weight-related comorbid condition receive ixekizumab and tirzepatide concomitantly administered, participants see improvement in their psoriasis and achieve weight reduction compared to when receiving ixekizumab.

Participation in this study includes up to 12 visits and could last up to 61 weeks including screening, open label treatment period, and post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate-to-severe plaque psoriasis (PsO) for at least 6 months.
* Have both a Static Physician's Global Assessment (sPGA) score of ≥3 and a Psoriasis Area and Severity Index (PASI) ≥12.
* Have ≥10% body surface area (BSA) involvement.
* Have obesity, body mass index of ≥30 kilograms per meter squared (BMI ≥30 kg/m²) or overweight (BMI ≥27 to <30 kg/m²) in the presence of at least 1 of these weight-related comorbid conditions (hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease, or T2DM).

Exclusion Criteria:

Medical Conditions

* Have Type 1 Diabetes Mellitus (T1DM).
* Have insulin-treated Type 2 Diabetes Mellitus (T2DM).
* Have a prior or planned surgical treatment for obesity.
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia (MEN) syndrome type 2.
* Have active, or a history of inflammatory bowel disease (Crohn's or ulcerative colitis).
* Have a diagnosis or history of malignant disease within the 5 years prior to randomization, with the following exceptions:

  * basal cell or squamous epithelial carcinomas of the skin that have been resected, with no evidence of metastatic disease for 3 years.
  * cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to randomization.
* Have serious disorder or illness other than PsO.
* Have a history of chronic or acute pancreatitis.
* Have any prior use of ixekizumab or tirzepatide.
* Have a previous failure or intolerance to an interleukin 17 inhibitor (IL-17i) or glucagon-like peptide 1 (GLP-1) receptor agonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Simultaneously Achieved Psoriasis Area and Severity Index (PASI) 100 and At Least 10% Weight Reduction | Baseline to Week 36
  PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (none) to 4 (very severe). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no psoriasis) to 72 (the most severe disease).Participants achieving PASI 100 were defined as having an improvement of at least 100% in the PASI score compared to baseline.

SECONDARY OUTCOMES:
Percentage of Participants Who Simultaneously Achieved PASI 75 and At Least 5% Weight Reduction | Baseline to Week 36
  PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (none) to 4 (very severe). Each area is scored separately, and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no psoriasis) to 72 (the most severe disease). Participants achieving PASI 75 were defined as having an improvement of ≥75% in the PASI score compared to baseline.
Percentage of Participants Achieving PASI 100 | Baseline to Week 36
  PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (none) to 4 (very severe). Each area is scored separately, and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no psoriasis) to 72 (the most severe disease). Participants achieving PASI 100 were defined as having an improvement of at least 100% in the PASI scores compared to baseline.
Percentage of Participants Achieving At Least 10% Weight Reduction | Baseline to Week 36
  Percentage of Participants Who Achieved at Least a 10% Weight Reduction

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (72):
- United States (68):
  - Total Skin & Beauty Dermatology Center, PC DBA Total Dermatology, Birmingham, Alabama
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Yuma Clinical Trials, Yuma, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Avance Clinical Trials, Laguna Niguel, California
  - Metropolis Dermatology, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - Cura Clinical Research - Oxnard, Oxnard, California
  - Integrative Skin Science and Research - Location 2, Sacramento, California
  - Therapeutics Clinical Research, San Diego, California
  - Life Clinical Trials, Coral Springs, Florida
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - NeoClinical Research, Hialeah, Florida
  - Skin Care Research, Hollywood, Florida
  - Encore Medical Research, Hollywood, Florida
  - Solutions Through Advanced Research, Jacksonville, Florida
  - Deluxe Health Center, Miami Lakes, Florida
  - Renstar Medical Research, Ocala, Florida
  - Leading Edge Dermatology, Plantation, Florida
  - International Clinical Research - Sanford, Sanford, Florida
  - Nodal Medical Center, Tampa, Florida
  - Palm Harbor Dermatology PA d/b/a TrueBlue Clinical Research, Tampa, Florida
  - DeNova Research, Chicago, Illinois
  - Oak Dermatology, Naperville, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Equity Medical - Bowling Green, Bowling Green, Kentucky
  - DelRicht Research, Baton Rouge, Louisiana
  - Care Access - Lake Charles (Bayou Pines), Lake Charles, Louisiana
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - Lawrence J. Green, MD, LLC, Rockville, Maryland
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - The Derm Institute of West Michigan, Caledonia, Michigan
  - MI Skin Innovations, Northville, Michigan
  - Las Vegas Dermatology, Las Vegas, Nevada
  - Skin Cancer and Dermatology Institute - Reno, Reno, Nevada
  - ActivMed Practices & Research, LLC., Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Care Access - Hoboken, Hoboken, New Jersey
  - Equity Medical, New York, New York
  - Mount Sinai Doctors - East 85th Street, New York, New York
  - Onsite Clinical Solutions - Huntersville, Huntersville, North Carolina
  - Red River Research Partners, Fargo, North Dakota
  - Optima Research - Boardman, Boardman, Ohio
  - Dermatologists of Southwest Ohio, Mason, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Columbia Dermatology & Aesthetics, Columbia, South Carolina
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - DelRicht Research - Thompson's Station, Smyrna, Tennessee
  - Tekton Research - Westlake Drive, Austin, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Tanner Clinic, Layton, Utah
  - Care Access - Arlington, Arlington, Virginia
  - Care Access - Danville, Danville, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Bellevue Dermatology Clinic, Bellevue, Washington
  - Dermatology of Seattle, Burien, Washington
- Puerto Rico (4):
  - SCB Research Center, Bayamón
  - Office of Dr. Alma M. Cruz, Carolina
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
  - Mindful Medical Research, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/